CLINICAL TRIAL: NCT02545361
Title: A Phase 1/2a, Multi-center, Dose Escalation, 2 Stages Study to Evaluate the Safety, Tolerability, and Anti-cancer Activity of Subcutaneously Administered KAHR-102 for the Treatment of Lymphoma Patients Who Express Both B7 and FasR
Brief Title: Safety, Tolerability, and Anti-cancer Activity of KAHR-102 (The Study Drug) for the Treatment of Lymphoma Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Program de-prioritized
Sponsor: Kahr Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KAHR002
Record Dates: First submitted 2015-08-04; First posted 2015-09-10 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KAHR002 (Experimental): premedication (20mg Dexamethasone (IV), 10mg Loratadine (P.O), and 1gr Paracetamol (P.O), 1 hour before treatment) with 2µg/kg KAHR-102 subcutaneous (SC) injection
  Interventions: Drug: KAHR-102

INTERVENTIONS:
Drug: KAHR-102 — KAHR-102 is a dual signaling protein (DSP).KAHR-102 will be administrated subcutaneously. In Stage 1A, 3 KAHR-102 SC injections will continue to be given every 14 days with an interval of 28 days after 1st cycle and 14 days after 2nd cycle and following cycles.
  In Stage 1B and Stage 2, subjects will be administered 3 KAHR-102 SC injections given every 7 days with an interval of 28 days after 1st cycle and 14 days after 2nd cycle and following cycles.
  Planned doses for stage 1:
  Cohort A: 2µg/kg Cohort B: 4 µg/kg Cohort C: 8 µg/kg Cohort D: 12 µg/kg Each cohort will only begin its first administration of KAHR-102 SC injection when the cohort preceding it will not meet criteria for a DLT (at least 7 days).

SUMMARY:
The purpose of this study is to evaluate the safety and to determine the Dose Limiting Toxicity (DLT) and the Maximal Tolerated Dose (MTD) of KAHR-102.

DETAILED DESCRIPTION:
Subjects will have a screening visit for determination of eligibility. Up to 40 evaluable subjects will be included in the study; up to 30 in stage 1, and 10 in stage 2.

The study is divided into 2 stages:

* Dose escalation - Stage 1A and 1B
* Dose Confirmation Phase - Stage 2

Stage 1A:

Will start with 3 subjects receiving premedication (20mg Dexamethasone Intravenous (IV), 10mg Loratadine Per Os (P.O), and 1gr Paracetamol (P.O), 1 hour before treatment) with 2 micrograms/kilograms (µg/kg) KAHR-102 subcutaneous (SC) injection every 14 days for 3 injections. 3 injections will be defined as 1 cycle.

Eligible subjects will be hospitalized for 48 hours following each study drug administration. Blood will be collected before and 24 hours (h) following the study drug administration for biochemistry, hematology and cytokine levels.

Pharmacokinetic (PK) samples will be collected during hospitalization for the first and third KAHR-102 SC injections. Sampling for PK will be repeated on Day 4, 7, 32 and 35.

Sampling for Anti Drug Antibodies (ADAs) will be taken before all 3 KAHR-102 SC injections. CT scan and ADAs will be repeated at Day 49.

Stage 1B:

Based on safety results from Stage 1A and Clinical Safety Committee (CSC) decision, 12 further eligible subjects will be assigned to 1 of 4 cohorts to receive a SC injection of KAHR-102 with pre-medication (20mg Dexamethasone (IV), 10mg Loratadine (P.O), and 1gr Paracetamol (P.O), all 1 hour before the KAHR-102 SC injection, once every 7 days for 3 injections starting with 2µg/kg KAHR-102 SC injection. 3 injections will be defined as 1 Cycle.

Eligible subjects will be hospitalized for 48 hours following each KAHR-102 SC injection.

Blood samples will be collected before and 24h following the administration of KAHR-102 SC injection for biochemistry, hematology and cytokines level.

PK samples will be collected during hospitalization for first and third KAHR-102 SC injections. PK will also be assessed on Days 4, 7 (before administration of second KAHR-102 SC injection), 18 and 21.

Sampling for ADA testing will be taken before administration of first and third KAHR-102 SC injections. CT scan and ADA sampling will be performed on Day 35.

Stage 2:

Following completion of Stage 1, safety assessment by CSC and determination of MTD will be performed. 10 subjects will be treated at MTD. KAHR-102 SC injection will be given every 7 days for 3 injections. 3 injections will be defined as 1 Cycle.

Subjects will be hospitalized during treatment for 48 hours following each KAHR-102 SC injection.

Blood will be collected before and 24h following the administration of KAHR-102 SC injection for biochemistry, hematology, cytokines level.

PK sampling will be taken during hospitalization for first and third KAHR-102 SC injections and repeated on days 4, 7(before administration of second injection), 18, 21.

Samples for ADA testing will be collected prior to the first and third KAHR-102 SC injections. At Day 35 ADA sampling and CT scan will be repeated.

Cycles will be repeated at a frequency of 28 days after third KAHR-102 SC injection of 1st cycle and 14 days after 2nd cycle and following cycles Treatment will be discontinued based on investigator decision if CT scan shows evidence of disease progression or for any safety issues. The process will be overseen by the CSC.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with recurrent malignant lymphoma, which express B7 and FasR and have either failed to respond to standard therapy, relapsed and for whom no standard therapy is available.
* Measurable disease as measured by "Lugano" Classification.
* A measurable node must have a longest diameter (LDi) greater than 1.5 cm. Measurable extranodal disease (eg, hepatic nodules) may be included in the six representative, measured lesions. A measurable extranodal lesion should have an LDi greater than 1.0 cm
* Biopsy of tumor stains positive to cluster of differentiation 95 (CD95) and to Cluster of Differentiation 80 (CD80) or Cluster of Differentiation 86 (CD86) or both within the last 6 months.
* If greater than 6 months , a fine-needle aspiration (FNA) should be performed
* Men and Women age > 18.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 3.
* Estimated life expectancy of at least 2 months.
* Adequate liver function (serum bilirubin ≤2.0 mg/100 ml; alanine aminotransferase, aspartate aminotransferase ≤2× ULN).
* Adequate renal function (serum creatinine ≤1.5 mg/100 ml or creatinine clearance ≥30 ml/min/1.73m2 as measured by Cockcroft -Gault / CKD (Chronic Kidney Disease)/EPI (Epidemiology Collaboration) formulas.
* Platelet count ≥ 50,000 and an absolute neutrophil count (ANC) ≥ 1500 /mm3.
* Women of child bearing potential practicing an acceptable method of birth control.
* Understanding of study procedures and willingness to comply for the entire length of the study and to give written informed consent.

Exclusion Criteria:

* Other standard anti-neoplastic therapies are available.
* Known Central Nervous System (CNS) lymphoma.
* Chronic lymphocytic leukemia and autoimmunity leukemia.
* Known hypersensitivity to the study drug or to any of its components.
* Chronic heat failure (CHF) New-York heart association (NYHA) = Class IV.
* Known Chronic Obstructive Pulmonary Disease (COPD) > Stage 3 (Forced Expiratory Volume -(FEV1)<50%, FEV1/Forced Vital Capacity (FVC)<70%).
* Chronic kidney disease (CKD) >Stage 4 (subjects with known Filtration rate (FR)<30 milliliter (mL)/min/1.73m2).
* Cirrhosis (Child-Pugh Class C score).
* Known hypersensitivity to drug components.
* Prior chemotherapy within 3 weeks, nitrosureas within 6 weeks, therapeutic anticancer antibodies within 3 weeks, radio or toxin immunoconjugates within 10 weeks, radiation therapy within 3 weeks, or major surgery within 28 days of first dose of the study drug.
* American Society for Cytotechnology (ASCT) and prior allogeneic stem cell transplantation (SCT)< 12 weeks prior to first dose of the study drug.
* Myelosuppressive treatment within 2-3 weeks of entering this study. Prednisone allowed.
* Any other severe concurrent disease which in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Positive test for acquired immune deficiency syndrome (AIDS).
* Any positive test for hepatitis B or hepatitis C virus (HBV or HCV) indicating acute or chronic infection (HBsAg, HBcAb total and anti-HCV Abs).
* Presence of uncontrolled infection.
* Evidence of active bleeding or bleeding susceptibility or medically significant hemorrhage within prior 30 days.
* Coumadin therapy.
* Pregnant or lactating.
* Treatment with other investigational drugs within 14 days of start of this study.
* Prisoners or subjects who are involuntarily incarcerated.
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate incidence of adverse events | Up to 9 months
  Safety, as determined by frequency, nature, and severity of adverse events; and the profile of dose limiting toxicities.

SECONDARY OUTCOMES:
Blood samplings for KAHR-102 levels | Stage 1A: Pre-dose, days 1, 2, 28, 29 (Injections 1 and 3). Stages 1B and 2: Pre-dose, days 1, 2 ,14 ,15 (Injections 1 and 3). Repeated on Day 4, 7, 32 and 35.
  KAHR-102 pharmacokinetic profile by plasma concentrations.
Blood sampling for Anti-Drug Antibodies (ADAs) | Stage 1A: Pre-dose day 1, 14, 28 in all cycles, day 49; Stages 1B and 2: Pre-dose day 1 and 28 in all cycles, day 35.
  Sampling for Anti-Drug Antibodies
Tumors measurements | Stage 1A: Pre-dose, day 49; Stages 1B and 2: Pre-dose, day 35 and every 10 weeks on average.
  CT scan
Optional "LUGANO" classification response | Stage 1A: Pre-dose, day 49; Stages 1B and 2: Pre-dose, day 35 and every 10 weeks on average.
  Evaluation, staging, and assessment of response in patients with Hodgkin lymphoma and non-Hodgkin lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Chava Sarfati, Pharm, Study Chair — Kahr Medical